CLINICAL TRIAL: NCT03655977
Title: Radiation Therapy Planning by Multi-parametric PET/MRI Imaging in Patients With Cervical Cancer
Acronym: RaPiCCa
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Rigshospitalet, Denmark (Other)
Responsible Party: Principal Investigator, heidi ryssel, medical doctor, Rigshospitalet, Denmark
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: H-17016438
Record Dates: First submitted 2018-08-02; First posted 2018-09-04 (Actual); Last update posted 2018-09-04 (Actual); Status verified 2018-08

CONDITIONS: Cervical Cancer
Keywords: Cervical cancer; Treatment planning; PET/MRI imaging
MeSH Terms: conditions — Uterine Cervical Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Cervical cancer patients (Experimental): This pilot study includes 25 women with histologically proven advanced stage primary cervical cancer (FIGO stages ≥IB2-IVA), planned for treatment with radio-chemotherapy.
  Interventions: Drug: 68Ga-NODAGA-E[c(RGDyK)]2; Device: PET/MRI scan instead of only MRI

INTERVENTIONS:
Drug: 68Ga-NODAGA-E[c(RGDyK)]2 — 200 MBq 68Ga-NODAGA-E[c(RGDyK)]2 will be administered before external beam radiation therapy (EBRT).
  Other Names: RGD-PET
Device: PET/MRI scan instead of only MRI — Following injection of RGD-PET the patients will be subjected to PET/MRI of the pelvic for planning external beam radiation therapy.
Drug: 68Ga-NODAGA-E[c(RGDyK)]2 — 200 MBq 68Ga-NODAGA-E[c(RGDyK)]2 will be administered before brachytherapy (BT).
  Other Names: RGD-PET
Device: PET/MRI scan instead of only MRI — Following injection of RGD-PET the patients will be subjected to PET/MRI of the pelvic for planning brachytherapy.

SUMMARY:
The main goal of this project is to evaluate the potential and feasibility of hybrid PET/MRI functional imaging to non-invasively measure tumor characteristics for radiation therapy planning (RT) for cervical cancer. It will be assessed how the complementary information of tumor characteristics can contributed to better understanding of tumor delineation. Another endpoint of this study is to evaluate a new PET-tracer (68Ga-NODAGA- E[c(RGDyK)]2) enabling imaging of tumor-angiogenesis.

DETAILED DESCRIPTION:
The standard treatment for patients with locally advanced cervical cancer includes a combination of external beam radiotherapy (EBRT) and brachytherapy (BT) with concurrent cisplatin-based chemotherapy. During the last decade, the utilization of MRI for planning of EBRT and BT has grown based on the GEC ESTRO recommendations and the cervix is among the first cancer sites where response-adaptive radiotherapy has been successfully implemented in clinical practice. This approach has changed patterns of clinical practice with regard to dose administration, and significant improvements in clinical outcome have been reported. However further development of both BT and EBRT is still demanded to improve tumor delineation and consequently local control.

Recent developments in advanced image guidance for both EBRT and BT have potential to improve local as well as nodal and also systemic control. Multi-parametric PET/MR imaging potentially offers new possibilities for RT planning, whereas a complete replacement of the planning MRI with combined PET/MRI for EBRT and BT, alters target volume delineation due to superior soft tissue contrast provided by MRI and combined with the information of tumor heterogeneity, perfusion characteristics, and hypoxia provided by PET, DW-MRI, and DCE-MRI. However combined use of PET/MRI for treatment planning still remains challenging due to several aspects. Therefore, investigators intend to encounter the technical challenges regarding dose planning and attenuation correction of MRI hardware and immobilization devices by generating Pseudo-CT, using methods based on ultra-short echo time (UTE) MR sequence. Additionally, investigators desire to assess how the complementary information provided by multi-parametric PET/MRI can affect the planning of EBRT and BT and contribute to better understanding of the pathology of cervical cancer during chemo-radiotherapy and improve radiation treatment.

The PET/MR will be performed with a new PET-tracer "RGD" (68Ga-NODAGA- E[c(RGDyK)]2) enabling imaging of tumor-angiogenesis. This is to show the angiogenesis within the tumor and changes during external radiotherapy. The study of angiogenesis will be supported by examination of tissues from the tumor.

Investigators expect the angiogenesis to correlate to the aggression and thereby the prognosis of the individual tumor.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with cervical cancer stage
* Tumor > 1cm
* Referred for EBRT and BT planning
* Age > 18 years
* Informed consent

Exclusion Criteria:

* Prior RT of the pelvic region
* Pregnancy and lactation
* Claustrophobia
* MR-incompatible implants

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2018-09-01 (Estimated); Primary Completion 2021-09-01 (Estimated); Study Completion 2021-09-01 (Estimated)

PRIMARY OUTCOMES:
Feasibility of PET/MRI in radiation treatment planning workflow | 1 year
  Assess the feasibility of PET/MRI in the radiation treatment planning workflow with respect to the adequacy of tumor delineation and planning target volume using PET/MRI data as compared to MRI-only planning.
Measure of angiogenesis with 68Ga-NODAGA-E[c(RGDyK)]2 radio-tracer in patient with cervical cancer | 1 hour
  Measure of voxel values, metabolic volume represents angiogenesis volume in patients with cervical cancer. Angiogenesis can be analysed qualitatively.

SECONDARY OUTCOMES:
Feasibility of dose planning using MRI | 1 year
  evaluate the feasibility of performing dose planning based on MRI-only obtained from a PET/MRI system by applying new sequence.
Changes in PTV between conventional MRI and PET/MRI | 1 month
  Compare changes in planning target volume (PTV) and tumor delineation between conventional MRI and PET/ MRI planning.
measuring tumor metabolism using Standard Uptake Value (SUV). | 1 hour
  Tumor metabolism in cancer cells prior to external beam radiation therapy as well as brachytherapy can be measured by SUV which depends on patient weight and injected activity.

CONTACTS AND LOCATIONS:
Overall Officials: Barbara Malene Fisher, Study Director — Dept. of Clinical Physiology, Nuclear Medicine and PET, Rigshospitalet
Locations (1):
- University Copenhagen, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: Undecided